CLINICAL TRIAL: NCT01220128
Title: Study of GSK2302024A Antigen-Specific Cancer Immunotherapeutic Combined With Standard Neoadjuvant Treatment in Patients With WT1-positive Primary Invasive Breast Cancer
Brief Title: Evaluation of an Anti-cancer Immunotherapy Combined With Standard Neoadjuvant Treatment in Patients With WT1-positive Primary Invasive Breast Cancer
Acronym: INDUCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study termination due to negative Ph III of another study product from same technology platform.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 113172; 2010-019909-42 (EudraCT Number)
Record Dates: First submitted 2010-10-07; First posted 2010-10-13 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-04

CONDITIONS: Neoplasms, Breast
Keywords: WT1; neoadjuvant; tumor antigen; immunotherapy; breast cancer; adult
MeSH Terms: conditions — Breast Neoplasms | interventions — Aromatase Inhibitors; Fluorouracil; Cyclophosphamide; Docetaxel; Doxorubicin; Epirubicin; Paclitaxel; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (7):
- Cohort A-GSK2302024A Group (Experimental): This group included postmenopausal patients with hormone receptor-positive breast cancer who received aromatase inhibitor (AI) as neoadjuvant therapy, concurrently with administration of GSK2302024A according to the treatment schedule.
  Interventions: Biological: GSK Biologicals' recombinant WT1 Antigen-Specific Cancer Immunotherapeutic (ASCI) GSK2302024A; Drug: Aromatase inhibitor
- Cohort A-Placebo Group (Placebo Comparator): This group included postmenopausal patients with hormone receptor-positive breast cancer who received aromatase inhibitor (AI) as neoadjuvant therapy, concurrently with administration of placebo, according to the treatment schedule.
  Interventions: Drug: Placebo; Drug: Aromatase inhibitor; Drug: 5-Fluorouracil; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin; Drug: Epirubicin; Drug: Paclitaxel
- Cohort B-GSK2302024A Group (Experimental): This group included breast cancer patients who received GSK2302024A, 5-Fluorouracil, Cyclophosphamide, Docetaxel, Doxorubicin, Epirubicin and Paclitaxel according to the treatment schedule.
  Interventions: Biological: GSK Biologicals' recombinant WT1 Antigen-Specific Cancer Immunotherapeutic (ASCI) GSK2302024A; Drug: 5-Fluorouracil; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin; Drug: Epirubicin; Drug: Paclitaxel
- Cohort B-Placebo Group (Placebo Comparator): This group included breast cancer patients who received placebo, 5-Fluorouracil, Cyclophosphamide, Docetaxel, Doxorubicin, Epirubicin and Paclitaxel according to the treatment schedule.
  Interventions: Drug: Placebo; Drug: 5-Fluorouracil; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin; Drug: Epirubicin; Drug: Paclitaxel
- Cohort C-GSK2302024A Group (Experimental): This group included patients with Human Epidermal Growth Factor Receptor 2 (HER2)-overexpressing breast cancer who received neoadjuvant trastuzumab (Herceptin) therapy, concurrently with administration of GSK2302024A, 5-Fluorouracil, Carboplatin, Cyclophosphamide, Docetaxel, Doxorubicin, Epirubicin and Paclitaxel according to the treatment schedule.
  Interventions: Biological: GSK Biologicals' recombinant WT1 Antigen-Specific Cancer Immunotherapeutic (ASCI) GSK2302024A; Drug: 5-Fluorouracil; Drug: Carboplatin AUC; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin; Drug: Epirubicin; Drug: Paclitaxel; Drug: Trastuzumab
- Cohort C-Placebo Group (Placebo Comparator): This group included patients with Human Epidermal Growth Factor Receptor 2 (HER2)-overexpressing breast cancer who received neoadjuvant trastuzumab (Herceptin) therapy, concurrently with administration of placebo, 5-Fluorouracil, Carboplatin, Cyclophosphamide, Docetaxel, Doxorubicin, Epirubicin and Paclitaxel according to the treatment schedule.
  Interventions: Drug: Placebo; Drug: 5-Fluorouracil; Drug: Carboplatin AUC; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin; Drug: Epirubicin; Drug: Paclitaxel; Drug: Trastuzumab
- Cohort D-GSK2302024A-D14 Group (Experimental): This group included patients with hormone receptor-positive and HER2 non-overexpressing breast cancer, who received GSK2302024A, 5-Fluorouracil, Cyclophosphamide, Docetaxel, Doxorubicin, Epirubicin and Paclitaxel according to the treatment schedule.
  Interventions: Biological: GSK Biologicals' recombinant WT1 Antigen-Specific Cancer Immunotherapeutic (ASCI) GSK2302024A; Drug: 5-Fluorouracil; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin; Drug: Epirubicin; Drug: Paclitaxel

INTERVENTIONS:
Biological: GSK Biologicals' recombinant WT1 Antigen-Specific Cancer Immunotherapeutic (ASCI) GSK2302024A — 6 or 8 injections at 3 weeks apart, injected intramuscularly in the deltoid or lateral region of the thigh.
  Other Names: WT1 ASCI
  Arms: Cohort A-GSK2302024A Group; Cohort B-GSK2302024A Group; Cohort C-GSK2302024A Group; Cohort D-GSK2302024A-D14 Group
Drug: Placebo — 6 or 8 doses at 3 weeks apart of sucrose/mannitol-based formulation reconstituted with an oil-in-water emulsion, injected intramuscularly in the deltoid or lateral region of the thigh.
  Arms: Cohort A-Placebo Group; Cohort B-Placebo Group; Cohort C-Placebo Group
Drug: Aromatase inhibitor — This treatment consisted of any aromatase inhibitor (e.g. letrozole or exemestane), administered intravenously in Cohort A Groups daily for either 18 (if 6 doses of WT1 ASCI/placebo) or 24 weeks (if 8 doses of WT1 ASCI/placebo).
  Arms: Cohort A-GSK2302024A Group; Cohort A-Placebo Group
Drug: 5-Fluorouracil — Administered intravenously in Cohorts A Placebo, B, C and D/E Groups: for the 6 WT1 ASCI-dose schedule 3 doses at 3 weeks apart, and for the 8 WT1 ASCI-dose schedule 4 doses at 3 weeks apart. For Cohorts A Placebo, B and C Groups, the administration was on the same day as the administration of WT1 ASCI/placebo (Day 1 of each cycle). For Cohort D/E Groups, the administration was on Day 14 of each cycle.
  Arms: Cohort A-Placebo Group; Cohort B-GSK2302024A Group; Cohort B-Placebo Group; Cohort C-GSK2302024A Group; Cohort C-Placebo Group; Cohort D-GSK2302024A-D14 Group
Drug: Carboplatin AUC — Administered intravenously in Cohort C Groups in 6 doses at 3 weeks apart, on the same day as WT1 ASCI/placebo administration (Day 1 of each cycle).
  Arms: Cohort C-GSK2302024A Group; Cohort C-Placebo Group
Drug: Cyclophosphamide — Administered intravenously in Cohorts A Placebo, B, C and D/E Groups: for the 6 WT1 ASCI-dose schedule 3 doses in Cohort C Groups and 6 doses 3 weeks apart in Cohorts A Placebo, B and D Groups, while for the 8 WT1 ASCI-dose schedule 4 doses at 3 weeks apart. For Cohorts A Placebo, B and C Groups, the administration was on the same day as the administration of WT1 ASCI/placebo (Day 1 of each cycle). For Cohort D/E Groups, the administration was on Day 14 of each cycle.
  Arms: Cohort A-Placebo Group; Cohort B-GSK2302024A Group; Cohort B-Placebo Group; Cohort C-GSK2302024A Group; Cohort C-Placebo Group; Cohort D-GSK2302024A-D14 Group
Drug: Docetaxel — Administered intravenously in Cohorts A Placebo, B, C and D/E Groups: for the 6 WT1 ASCI-dose schedule 3 or 6 doses 3 weeks apart, while for the 8 WT1 ASCI-dose schedule 4 doses at 3 weeks apart. For Cohorts A Placebo, B and C Groups, the administration was on the same day as the administration of WT1 ASCI/placebo (Day 1 of each cycle). For Cohort D/E Groups, the administration was on Day 14 of each cycle.
  Arms: Cohort A-Placebo Group; Cohort B-GSK2302024A Group; Cohort B-Placebo Group; Cohort C-GSK2302024A Group; Cohort C-Placebo Group; Cohort D-GSK2302024A-D14 Group
Drug: Doxorubicin — Administered intravenously in Cohorts A Placebo, B, C and D/E Groups: for the 6 WT1 ASCI-dose schedule 6 doses 3 weeks apart (Cohort C patients with this schedule did not receive this treatment), while for the 8 WT1 ASCI-dose schedule 4 doses at 3 weeks apart. For Cohorts A Placebo, B and C Groups, the administration was on the same day as the administration of WT1 ASCI/placebo (Day 1 of each cycle). For Cohort D/E Groups, the administration was on Day 14 of each cycle.
  Arms: Cohort A-Placebo Group; Cohort B-GSK2302024A Group; Cohort B-Placebo Group; Cohort C-GSK2302024A Group; Cohort C-Placebo Group; Cohort D-GSK2302024A-D14 Group
Drug: Epirubicin — Administered intravenously in Cohorts A Placebo, B, C and D/E Groups: for the 6 WT1 ASCI-dose schedule 3 doses 3 weeks apart, while for the 8 WT1 ASCI-dose schedule 4 doses at 3 weeks apart. For Cohorts A Placebo, B and C Groups, the administration was on the same day as the administration of WT1 ASCI/placebo (Day 1 of each cycle). For Cohort D/E Groups, the administration was on Day 14 of each cycle.
  Arms: Cohort A-Placebo Group; Cohort B-GSK2302024A Group; Cohort B-Placebo Group; Cohort C-GSK2302024A Group; Cohort C-Placebo Group; Cohort D-GSK2302024A-D14 Group
Drug: Paclitaxel — Administered intravenously in Cohorts A Placebo, B, C and D/E Groups: only in the 8 WT1 ASCI-dose schedule patients received 4 at 3 weeks apart or 12 weekly doses. For Cohorts A Placebo, B and C Groups, the administration was on the same day as the administration of WT1 ASCI/placebo (Day 1 of each cycle). For Cohort D/E Groups, the administration was on Day 14 of each cycle.
  Arms: Cohort A-Placebo Group; Cohort B-GSK2302024A Group; Cohort B-Placebo Group; Cohort C-GSK2302024A Group; Cohort C-Placebo Group; Cohort D-GSK2302024A-D14 Group
Drug: Trastuzumab — Administered intravenously in Cohort C Groups: for the 6 WT1 ASCI-dose schedule 3 or 6 doses 3 weeks apart, while for the 8 WT1 ASCI-dose schedule 4 doses at 3 weeks apart. For Cohort B and C Groups, the administration was on the same day as the administration of WT1 ASCI/placebo (Day 1 of each cycle). For Cohort D/E Groups, the administration was on Day 14 of each cycle.
  Arms: Cohort C-GSK2302024A Group; Cohort C-Placebo Group

SUMMARY:
The purpose of this study is to evaluate the safety, immunogenicity and clinical activity of a new WT1 anti-cancer immunotherapy in patients with WT1-positive Stage II or III breast cancer. The treatment will be given before surgery in combination with standard therapy.

DETAILED DESCRIPTION:
The study will be conducted in two consecutive segments (Phase I and Phase II), each with specific objectives. Active follow-up will be for three years.

Patients in this study will be allocated to cohorts as below. Cohort A will include postmenopausal patients with hormone receptor-positive breast cancer who receive aromatase inhibitor (AI) as neoadjuvant therapy concurrently with administration of 6 or 8 doses of WT1 anti-cancer immunotherapy (WT1 ASCI)/placebo starting on Day 0. AI treatment will be administered daily for duration of either 18 (if 6 doses of WT1 ASCI/placebo) or 24 weeks (if 8 doses of WT1 ASCI/placebo).

Cohort B will include breast cancer patients who will receive neoadjuvant chemotherapy concurrently with administration of WT1 ASCI/placebo starting on Day 0. Neoadjuvant chemotherapy in Cohort B will consist either 1) if 6 doses of WT1 ASCI/placebo: 6 cycle-treatment chemotherapy regimens consist of 6, three-weekly cycles of anthracycline/taxane-based therapy, or 2) if 8 doses of WT1 ASCI/placebo: 8 cycle-treatment regimens consisting of 4 three-weekly cycles of anthracycline-based therapy followed by 4 three-weekly or 12-weekly taxane administrations without trastuzumab.

Cohort C will include patients with Human Epidermal Growth Factor Receptor 2 (HER2)-overexpressing breast cancer who will receive neoadjuvant trastuzumab (Herceptin) therapy combined with chemotherapy concurrently with administration of WT1 ASCI/placebo starting on Day 0. Neoadjuvant chemotherapy in Cohort C will consist either 1) if 6 doses of WT1 ASCI/placebo: 6 cycle-treatment chemotherapy regimens consist of 6, three-weekly cycles of anthracycline/taxane-based therapy, or 2) if 8 doses of WT1 ASCI/placebo: 8 cycle-treatment regimens consisting of 4 three-weekly cycles of anthracycline-based therapy followed by 4 three-weekly or 12-weekly taxane administrations with trastuzumab.

Cohorts D and E will include patients with hormone receptor-positive and HER2 non-overexpressing breast cancer who will receive neoadjuvant chemotherapy. For patients in these Cohorts D and E, WT1 ASCI/placebo (placebo applicable only for Cohort E patients) will be administered on Day 14 of each three-weekly cycle of chemotherapy. Neoadjuvant chemotherapy in Cohorts D and E will consist either 1) if 6 doses of WT1 ASCI/placebo: 6 cycle-treatment chemotherapy regimens consist of 6, three-weekly cycles of anthracycline/taxane-based therapy, or 2) if 8 doses of WT1 ASCI/placebo: 8 cycle-treatment regimens consisting of 4 three-weekly cycles of anthracycline-based therapy followed by 4 three-weekly taxane administrations without trastuzumab. Enrolment in Cohort E will be conditional on the absence of a safety signal and on the adequate induction of an immune response by the WT1 ASCI in Cohort D (defined as >= 40% response rate based on post-Dose 4 anti-WT1 antibody responses in at least six patients). If this criterion is met, 60 patients (40 receiving WT1 ASCI and 20 placebo) with identical eligibility criteria will be enrolled into Cohort E. In case no adequate safety and/or immunogenicity will be obtained in Cohort D, recruitment in Cohort E will not be initiated.

The protocol has been updated following Protocol Amendment 4, April 2013, leading to the update of the study design.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥ 18 years of age at the time the informed consent to screening has been obtained.
* The patient has proven T1 with lymph node involvement or T2-T4c, any N, M0 primary invasive breast cancer, histologically confirmed by core needle biopsy.

Isolated supraclavicular lymph node involvement is allowed.

* The patient's tumor shows WT1 antigen expression.
* The patient has one of the following histologically confirmed breast cancer subtypes:

  * Estrogen receptor and/or progesterone positive tumor.
  * Human epidermal growth factor receptor 2 (HER2)-overexpressing breast cancer.
  * HER2-negative breast cancer.
* Eastern Cooperative Oncology Group (performance status of 0 or 1 at the time of study treatment allocation.
* Baseline left ventricular ejection fraction of ≥ 50% as measured within six weeks prior to study treatment allocation by echocardiography or multi-gated acquisition(MUGA)scan.
* The patient shows normal organ function according to the following parameters(as measured within six weeks prior to treatment allocation)::

  * Hemoglobin: Within normal range according to institutional standards.
  * Absolute leukocyte count: Within normal range according to institutional standards.
  * Absolute lymphocyte count: Within normal range according to institutional standards.
  * Platelet count: Within normal range according to institutional standards
  * Alanine aminotransferase: ≤ 2.5 x Upper Limit of Normal (ULN)
  * Aspartate aminotransferase: ≤ 2.5 x ULN
  * Total bilirubin: ≤ 1.5 x ULN. In the case of known Gilbert's syndrome ≤ 2 x ULN
  * Serum creatinine: 1.5 x ULN
  * Calculated creatinine clearance: > 50 mL/min
* A female patient of childbearing potential may be enrolled in the study, if the patient:

  * has practiced adequate contraception for 30 days prior to study product administration, and
  * has a negative pregnancy test within one week prior to treatment allocation and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the study product administration series.In view of the investigator, the patient can and will comply with the requirements of the protocol.
* Written informed consent has been obtained from the patient prior to performance of any study specific procedure.

Exclusion Criteria:

* The patient has inflammatory breast cancer, which is defined as clinically significant erythema of the breast and/or documented dermal lymphatic invasion.
* Diagnosis established by incisional biopsy.
* Prior and concomitant neoadjuvant anti-breast-cancer treatments such as chemotherapy, immunotherapy / biological response modifiers, endocrine therapy, and radiotherapy, unless authorized specifically by the protocol.
* The patient is known to be human immunodeficiency virus -positive.
* The patient has symptomatic autoimmune disease such as, but not limited to multiple sclerosis, lupus, and inflammatory bowel disease. Patients with vitiligo are not excluded.
* The patient is known to have difficult-to-control hypertension, coronary artery disease, arrhythmia requiring treatment, clinically significant valvular disease, cardiomegaly on chest X-ray, ventricular hypertrophy on electrocardiogram or previous myocardial infarction or congestive heart failure.
* The patient has a history of allergic reactions likely to be exacerbated by any component of the investigational product used in the study.
* The patient has other concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* The patient has (or has had) previous or concomitant malignancies at other sites, except effectively treated malignancy that is considered by the investigator highly likely to have been cured.
* The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent or to comply with the study procedures.
* The patient has received any investigational or non-registered product within 30 days preceding the first dose of study products or planned use during the study period.
* The patient requires concomitant treatment with any immunosuppressive agents or with systemic corticosteroids prescribed for chronic treatment.
* The patient has a significant disorder of coagulation or receives treatment with warfarin derivatives or heparin. Patients receiving individual doses of low molecular weight heparin outside of 24 hours prior to WT1-A10 + AS15 ASCI/placebo administration are eligible. Patients receiving prophylactic antiplatelet medications e.g. low-dose aspirin, and without a clinically-apparent bleeding tendency are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-04-11 (Actual); Primary Completion 2014-11-14 (Actual); Study Completion 2014-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (35):
- United States (8):
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Bend, Oregon
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Spokane, Washington
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Namur
- France (2):
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Saint-Herblain
- Germany (8):
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Kiel, Schleswig-Holstein
- Italy (7):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Aviano (PN), Friuli Venezia Giulia
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Trento, Trentino-Alto Adige
- Russia (2):
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
- United Kingdom (5):
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Bournemouth
  - GSK Investigational Site, Derby
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site (click on the link provided below).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=19610

REFERENCES:
- [Derived] Higgins M, Curigliano G, Dieras V, Kuemmel S, Kunz G, Fasching PA, Campone M, Bachelot T, Krivorotko P, Chan S, Ferro A, Schwartzberg L, Gillet M, De Sousa Alves PM, Wascotte V, Lehmann FF, Goss P. Safety and immunogenicity of neoadjuvant treatment using WT1-immunotherapeutic in combination with standard therapy in patients with WT1-positive Stage II/III breast cancer: a randomized Phase I study. Breast Cancer Res Treat. 2017 Apr;162(3):479-488. doi: 10.1007/s10549-017-4130-y. Epub 2017 Feb 7. PMID 28176175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 66 enrolled patients, 6 patients did not receive study product doses and were hence excluded prior to study start.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Cohort B-GSK2302024A Group: This group included breast cancer patients who received GSK2302024A, 5-Fluorouracil, Cyclophosphamide, Docetaxel, Doxorubicin, Epirubicin and Paclitaxel, according to the treatment schedule.
Period: Overall Study
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Started | 15 | 7 | 9 | 6 | 11 | 4 | 8
Completed | 11 | 6 | 6 | 6 | 11 | 4 | 3
Not Completed | 4 | 1 | 3 | 0 | 0 | 0 | 5
Not completed — Progressive disease | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Sponsor study termination | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse event, serious fatal | 2 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse event, non-fatal | 1 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Consent withdrawn by subject | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group | Total
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.3 (10.4) | 70.9 (7.1) | 49.3 (15.6) | 60.7 (9.8) | 52.9 (10.6) | 53.3 (6.2) | 49.6 (8.7) | 58.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 9 | 6 | 11 | 4 | 8 | 60
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Severe Toxicities
Description: Severe toxicity was defined as follows: - A Grade 3 or higher toxicity that is related or possibly related to the combined administration of standard treatment and GSK2302024A/placebo - A decrease in Left Ventricular Ejection Fraction (LVEF) from baseline with ≥ 10 points and at < 50% that is related or possibly related to the combined administration of treatment and that is confirmed by a second LVEF assessment within approximately 3 weeks. - A Grade 2 or higher cardiac ischemia/infarction that is related or possibly related to the combined administration of standard treatment and GSK2302024A /placebo. - A Grade 2 or higher allergic reaction occurring within 24 hours following the administration. - A Grade 3 or higher blood/bone marrow toxicity that was considered as related or possibly related to the combined Administration. - A decrease in renal function at the time of administration that was considered as related or possibly related.
Time Frame: From Week 0 to Week 26/32 (period starting from GSK2302024A/placebo treatment allocation and ending with the concluding Visit i.e.: Week 26 for patients receiving 6 injections and Week 32 for patients receiving 8 injections)
Population: The Total Treated Population included all patients who have received at least one dose of GSK2302024A study product or placebo.
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects | 0 | 0 | 1 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Patients With an Anti-Wilm's Tumor Gene (Anti-WT1) Humoral Response
Description: For initially seronegative patients: post-administration antibody concentration ≥ 9 EU/mL For initially seropositive patients: post-administration antibody concentration ≥ 2 fold the pre-administration antibody concentration.
Time Frame: At post-GSK2302024A/placebo Dose 4 (Week 13)
Population: According-to-Protocol (ATP) Population for immunogenicity included all eligible patients who did not report major protocol deviation, who had at least received the first 4 doses of study product and provided a valid result for immunogenicity measurement within the 4 weeks following Dose 4.
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 10 | 4 | 8 | 6 | 11 | 3 | 3
Subjects | 10 | 0 | 0 | 0 | 6 | 0 | 2

3. Primary Outcome: Number of Patients With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation patient, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse.
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects | 15 | 5 | 9 | 6 | 11 | 4 | 7

4. Primary Outcome: Number of Subjects With Serious Adverse Events SAE(s)
Description: A serious adverse event (SAE) is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of hospitalization, causes disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study patient. In this study, an event which was part of the natural course of the disease under study (i.e., disease progression/recurrence) was captured in the study/as an efficacy measure. Therefore it was not reported as an SAE. Progression/recurrence of the tumor was recorded in the clinical assessments in the electronic case report form (eCRF). Death due to progressive disease was recorded on a specific form in the eCRF but not as an SAE.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects | 3 | 0 | 4 | 2 | 5 | 1 | 5

5. Primary Outcome: Number of Subjects With Alanine Aminotransferase Increased Abnormality, by Common Terminology Criteria for Adverse Events (CTCAE) Maximum Grade
Description: Criteria for Adverse Events (CTCAE), version 4.0 of May 28, 2009. Grades refer to the severity of the AE: mild (grade 1), moderate (grade 2), severe or medically significant (grade 3), life-threatening (grade 4) and death (grade 5).
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 12 | 5 | 8 | 4 | 6 | 2 | 1
  Grade 1 | 2 | 1 | 1 | 2 | 5 | 2 | 2
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 1 | 1 | 0 | 0 | 0 | 0 | 5

6. Primary Outcome: Number of Subjects With Alkaline Phosphatase Increased Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 10 | 5 | 8 | 6 | 7 | 3 | 1
  Grade 1 | 5 | 1 | 1 | 0 | 4 | 1 | 2
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 5

7. Primary Outcome: Number of Subjects With Anemia, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 12 | 7 | 1 | 0 | 0 | 0 | 2
  Grade 1 | 2 | 0 | 7 | 4 | 7 | 3 | 2
  Grade 2 | 1 | 0 | 0 | 0 | 4 | 1 | 0
  Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 4

8. Primary Outcome: Number of Subjects With Aspartate Aminotransferase Increased Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 12 | 4 | 8 | 6 | 7 | 1 | 2
  Grade 1 | 3 | 2 | 1 | 0 | 4 | 3 | 1
  Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 5

9. Primary Outcome: Number of Subjects With Blood Bilirubin Increased Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 15 | 5 | 9 | 6 | 11 | 2 | 3
  Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 5

10. Primary Outcome: Number of Subjects With Creatine Increased Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 11 | 4 | 8 | 5 | 10 | 3 | 3
  Grade 1 | 4 | 2 | 1 | 1 | 1 | 1 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 4 | 1 | 0 | 0 | 0 | 0 | 5

11. Primary Outcome: Number of Subjects With Hemoglobin Increased Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 15 | 6 | 9 | 6 | 11 | 4 | 4
  Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 4

12. Primary Outcome: Number of Subjects With Hypercalcemia Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 14 | 3 | 8 | 6 | 11 | 4 | 3
  Grade 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 3 | 1 | 0 | 0 | 0 | 0 | 5

13. Primary Outcome: Number of Subjects With Hyperkalemia Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 15 | 5 | 7 | 6 | 10 | 4 | 3
  Grade 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
  Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 5

14. Primary Outcome: Number of Subjects With Hypernatremia Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 14 | 4 | 9 | 6 | 10 | 4 | 3
  Grade 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 5

15. Primary Outcome: Number of Subjects With Hypoalbuminemia Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 13 | 6 | 9 | 5 | 9 | 3 | 3
  Grade 1 | 1 | 0 | 0 | 1 | 2 | 1 | 0
  Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 5

16. Primary Outcome: Number of Subjects With Hypocalcemia Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 12 | 6 | 5 | 4 | 10 | 3 | 3
  Grade 1 | 3 | 0 | 3 | 1 | 1 | 1 | 0
  Grade 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 5

17. Primary Outcome: Number of Subjects With Hypokalemia Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 15 | 6 | 9 | 6 | 10 | 4 | 3
  Grade 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 5

18. Primary Outcome: Number of Subjects With Hyponatremia Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and post 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 15 | 6 | 5 | 6 | 11 | 4 | 3
  Grade 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 5

19. Primary Outcome: Number of Subjects With Lymphocyte Count Decreased Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 9 | 4 | 0 | 0 | 2 | 1 | 1
  Grade 1 | 5 | 2 | 3 | 2 | 3 | 1 | 1
  Grade 2 | 1 | 1 | 5 | 2 | 5 | 1 | 2
  Grade 3 | 0 | 0 | 1 | 2 | 1 | 1 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 4

20. Primary Outcome: Number of Subjects With Lymphocyte Count Increased Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 15 | 7 | 9 | 6 | 11 | 4 | 4
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 4

21. Primary Outcome: Number of Subjects With Neutrophil Count Decreased Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 12 | 6 | 7 | 5 | 10 | 3 | 0
  Grade 1 | 3 | 0 | 1 | 1 | 1 | 0 | 0
  Grade 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Grade Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 4

22. Primary Outcome: Number of Subjects With Platelet Count Decreased Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Grade 0 | 14 | 6 | 8 | 5 | 5 | 2 | 2
  Grade 1 | 1 | 1 | 1 | 1 | 5 | 2 | 2
  Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 4

23. Primary Outcome: Number of Subjects With White Blood Cell Decreased Abnormality, by CTCAE Maximum Grade
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 13 | 7 | 6 | 3 | 7 | 4 | 8
Subjects
  Grade 0 | 13 | 7 | 6 | 3 | 7 | 2 | 0
  Grade 1 | 2 | 0 | 2 | 2 | 4 | 1 | 1
  Grade 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 4

24. Primary Outcome: Number of Patients With Adverse Events (AEs), by CTCAE Maximum Grade Reported
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Any AE(s) Grade 1 | 6 | 1 | 0 | 0 | 0 | 0 | 0
  Any AE(s) Grade 2 | 6 | 4 | 6 | 0 | 4 | 3 | 2
  Any AE(s) Grade 3 | 3 | 0 | 0 | 5 | 3 | 0 | 1
  Any AE(s) Grade 4 | 0 | 0 | 2 | 1 | 4 | 1 | 4
  Any AE(s) Grade 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Any AE(s) | 15 | 5 | 9 | 6 | 11 | 4 | 7

25. Primary Outcome: Number of Subjects With Adverse Events (AEs) Assessed by the Investigators as Causally Related to GSK2302024A Treatment, by CTCAE Maximum Grade Reported
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Any related AE(s) Grade 1 | 7 | 2 | 0 | 0 | 5 | 0 | 2
  Any related AE(s) Grade 2 | 4 | 0 | 3 | 0 | 1 | 1 | 4
  Any related AE(s) Grade 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Any related AE(s) Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any related AE(s) Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any related AE(s) | 12 | 2 | 3 | 0 | 7 | 1 | 6

26. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs), by CTCAE Maximum Grade Reported
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Any SAE(s) Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE(s) Grade 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Any SAE(s) Grade 3 | 2 | 0 | 0 | 1 | 1 | 0 | 1
  Any SAE(s) Grade 4 | 0 | 0 | 2 | 1 | 4 | 1 | 4
  Any SAE(s) Grade 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Any SAE(s) | 3 | 0 | 4 | 2 | 5 | 1 | 5

27. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs), Assessed by the Investigators as Causally Related to GSK2302024A Treatment, by CTCAE Maximum Grade Reported
Description: as for outcome 5
Time Frame: During the treatment period and up to 30 days post last administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 15 | 7 | 9 | 6 | 11 | 4 | 8
Subjects
  Any related SAE(s) Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any related SAE(s) Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Any related SAE(s) Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Any related SAE(s) Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any related SAE(s) Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any related SAE(s) | 1 | 0 | 0 | 0 | 1 | 0 | 0

28. Primary Outcome: Number of Subjects With Breast Cancer Pathological Response
Description: The pathological response in lymph nodes was evaluated by presence or absence of tumor cells by histopathological examination. Partial responses mark the disappearance of tumor cells, with only small clusters or dispersed cells remaining (more than 90% loss) while complete response indicate no identifiable malignant cells. However, ductal carcinoma in situ may be present.
Time Frame: During the treatment period, up to Week 26/32
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
Number analyzed (Participants) | 13 | 6 | 9 | 6 | 11 | 4 | 4
Subjects
  Partial respose | 4 | 3 | 5 | 3 | 3 | 1 | 3
  Complete response | 0 | 0 | 0 | 2 | 6 | 3 | 1

ADVERSE EVENTS:
Time Frame: AEs were reported during the treatment period and up to 30 days post last administration. SAEs during the entire study period (Week 0 to Week 26/32).
Arm/Group | Cohort A-GSK2302024A Group | Cohort A-Placebo Group | Cohort B-GSK2302024A Group | Cohort B-Placebo Group | Cohort C-GSK2302024A Group | Cohort C-Placebo Group | Cohort D-GSK2302024A-D14 Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/7 | 1/9 | 0/6 | 0/11 | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/15 | 0/7 | 4/9 | 2/6 | 5/11 | 1/4 | 5/8
Other Adverse Events (participants affected / at risk) | 15/15 | 5/7 | 9/9 | 6/6 | 11/11 | 4/4 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A-GSK2302024A Group (N=15) | Cohort A-Placebo Group (N=7) | Cohort B-GSK2302024A Group (N=9) | Cohort B-Placebo Group (N=6) | Cohort C-GSK2302024A Group (N=11) | Cohort C-Placebo Group (N=4) | Cohort D-GSK2302024A-D14 Group (N=8)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A-GSK2302024A Group (N=15) | Cohort A-Placebo Group (N=7) | Cohort B-GSK2302024A Group (N=9) | Cohort B-Placebo Group (N=6) | Cohort C-GSK2302024A Group (N=11) | Cohort C-Placebo Group (N=4) | Cohort D-GSK2302024A-D14 Group (N=8)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 8 (8) | 4 (4) | 7 (7) | 4 (4) | 2 (2)
Injection site pain (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Injection site erythema (General disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 5 (5) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 6 (6) | 0 (0) | 8 (8) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 9 (9) | 5 (5) | 8 (8) | 3 (3) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.